CLINICAL TRIAL: NCT04982029
Title: Cannabidiol on reward-and Stress-related Neurocognitive Processes in Individuals With Opioid Use Disorder: A Double-blind, Placebo-controlled, Cross-over Trial
Brief Title: Cannabidiol on Reward- and Stress-related Neurocognitive Processes in Individuals With Opioid Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021P001829
Record Dates: First submitted 2021-06-19; First posted 2021-07-29 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: The study is a double-blind, placebo-controlled, cross-over trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double-blind cross-over trial, in which the research staff and participants will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol 600mg (Experimental): All subjects will receive 600mg of oral cannabidiol in a double-blind fashion. Cannabidiol will be provided using Epidiolex™ oral solution 100mg/mL. Following administration, a battery of tests will be conducted to examine reward- and stress-related neurocognitive processes.
  Interventions: Drug: Cannabidiol 100 MG/ML [Epidiolex]
- Placebo (Placebo Comparator): All subjects will receive a matching placebo in a double-blind fashion. Following administration, a battery of tests will be conducted to examine the impact on reward- and stress-related neurocognitive processes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol 100 MG/ML [Epidiolex] — 600mg
  Arms: Cannabidiol 600mg
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the impact of cannabidiol on reward- and stress-related neurocognitive processes among individuals with opioid use disorder on buprenorphine or methadone treatment.

DETAILED DESCRIPTION:
Individuals with opioid use disorder (OUD) demonstrate reward- and stress-related neurocognitive changes compared to individuals without OUD, including cravings for opioids in response to exposure to triggers, tendency to make impulsive and disadvantageous decisions, and a strong attentional bias towards drug-related cues. Together, these deficits are significant contributors to relapse and discontinuation of treatment. Cannabidiol (CBD) has been shown to impact some of these cognitive deficits but studies of CBD among individuals with OUD are mostly lacking. Therefore, this study aims to answer whether CBD has any impact on reward-related neurocognitive deficits in individuals with OUD. If successful, this line of research will lay the groundwork for future studies to evaluate CBD's impact on OUD treatment outcomes.

ELIGIBILITY:
Inclusion Criteria

* English speaking
* DSM5 diagnosis of opioid use disorder
* Receiving buprenorphine or methadone for treatment of opioid use disorder
* Agreeable to abstaining from using any cannabis or CBD products for the duration of the trial.

Exclusion Criteria:

* Any self-reported use of cannabis or CBD products in the past 30 days
* Baseline depression (PHQ9) or anxiety (GAD7) scores of greater than 10
* Currently pregnant
* Hepatic liver enzymes greater than 3x upper normal limit
* Hypersensitivity to cannabinoids or sesame oil (CBD solution comes in sesame oil emulsion)
* Currently taking any medications with known significant pharmacokinetic interactions with CBD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Rutland Medical Center, Rutland, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suzuki J, Prostko S, Szpak V, Chai PR, Spagnolo PA, Tenenbaum RE, Ahmed S, Weiss RD. Impact of cannabidiol on reward- and stress-related neurocognitive processes among individuals with opioid use disorder: A pilot, double-blind, placebo-controlled, randomized cross-over trial. Front Psychiatry. 2023 Mar 30;14:1155984. doi: 10.3389/fpsyt.2023.1155984. eCollection 2023. PMID 37065899

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study took place from April 2022 - December 2022 at Brigham and Women's Hospital in Boston and Rutland Medical Clinic in Rutland VT. Participants were recruited through clinics and patient registries.
Groups:
- Cannabidiol 600mg First, Placebo Second: In this condition, subjects will receive 600mg of oral cannabidiol in a double-blind fashion. Cannabidiol will be provided using Epidiolex™ oral solution 100mg/mL. Following administration, a battery of tests will be conducted to examine reward- and stress-related neurocognitive processes.
  Cannabidiol 100 MG/ML [Epidiolex]: 600mg
  In their second intervention visit, participants will receive a matched placebo. Following administration, a battery of tests will be conducted to examine reward- and stress-related neurocognitive processes.
  This group received CBD first and placebo second.
- Placebo First, Cannabidiol 600mg Second: Participants in this condition will receive a matched placebo in their first visit. Following administration, a battery of tests will be conducted to examine reward- and stress-related neurocognitive processes.
  In their second intervention visit, subjects will receive 600mg of oral cannabidiol in a double-blind fashion. Cannabidiol will be provided using Epidiolex™ oral solution 100mg/mL. Following administration, a battery of tests will be conducted to examine reward- and stress-related neurocognitive processes.
  Cannabidiol 100 MG/ML [Epidiolex]: 600mg
Period: Overall Study
Arm/Group | Cannabidiol 600mg First, Placebo Second | Placebo First, Cannabidiol 600mg Second
Started | 7 | 8
Baseline (This milestone represents the baseline measures and initial study visit.) | 7 | 8
First Intervention (This is the visit where participants receive their first intervention.) | 5 | 5
Second Intervention (This is the study visit where participants receive their second intervention after the 7-day washout period.) | 5 | 5
Completed | 5 | 5
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Cannabidiol 600mg First and Placebo Second: All subjects will receive 600mg of oral cannabidiol in a double-blind fashion. Cannabidiol will be provided using Epidiolex™ oral solution 100mg/mL. Following administration, a battery of tests will be conducted to examine reward- and stress-related neurocognitive processes.
  Cannabidiol 100 MG/ML [Epidiolex]: 600mg
  All subjects will receive a matching placebo in a double-blind fashion. Following administration, a battery of tests will be conducted to examine the impact on reward- and stress-related neurocognitive processes.
  Placebo: Matching placebo
  In this arm, participants received CBD first and placebo second.
- Placebo First and Cannabidiol 600mg Second: All subjects will receive 600mg of oral cannabidiol in a double-blind fashion. Cannabidiol will be provided using Epidiolex™ oral solution 100mg/mL. Following administration, a battery of tests will be conducted to examine reward- and stress-related neurocognitive processes.
  Cannabidiol 100 MG/ML [Epidiolex]: 600mg
  All subjects will receive a matching placebo in a double-blind fashion. Following administration, a battery of tests will be conducted to examine the impact on reward- and stress-related neurocognitive processes.
  Placebo: Matching placebo
  In this arm, participants received placebo first and CBD second.
- Not Randomized: In this condition, participants only completed the baseline visit and were lost to follow-up prior to randomization. Therefore, only baseline characteristics are reported for these individuals.
- Total: Total of all reporting groups
Arm/Group | Cannabidiol 600mg First and Placebo Second | Placebo First and Cannabidiol 600mg Second | Not Randomized | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (6.98) | 46 (11.40) | 33.6 (3.78) | 41.75 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 9
  Male | 1 | 3 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 4 | 5 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 5 | 5 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 15
Patient Health Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire (PHQ-9) is a questionnaire that quantifies depressive levels in participants. The PHQ-9 provides an assessment of depression severity. The minimum value is 0 and the maximum value is 27. Lower scores indicated lower levels of depression. The reliability, validity, and clinical utility of the PHQ-9 instrument are well-established.
  units on a scale | 7.2 (6.18) | 5.6 (2.61) | 10.4 (8.35) | 8.07 (6.17)
Generalized Anxiety Disorder 7 [Mean (Standard Deviation); unit: units on a scale] — The Generalized Anxiety Disorder 7 or the GAD7 is a questionnaire that measures anxiety in patients. It categorizes scores into mild, moderate and severe on a scale of 0-21, where lower scores represent more milder anxiety and higher scores more severe. Each individual question is a 4-point scale ranging 0 (none of the days) to 3 (almost all of the days).
  units on a scale | 9.2 (6.87) | 3.4 (3.21) | 10.2 (6.46) | 7.6 (6.16)
Brief Pain Inventory [Mean (Standard Deviation); unit: units on a scale] — The Brief Pain Inventory or BPI assesses severity of pain and impact on daily functioning. Higher BPI scores mean greater severity and impact on functioning and lower scores mean less severity and impact on functioning. Questions are on a scale of 0-10 and final scores are averages of questions.
  units on a scale
    Severity | 3 (2.5) | 3.8 (2.69) | 1.95 (1.87) | 2.82 (2.97)
    Interference | 3.51 (3.57) | 3.2 (3.28) | 3.69 (3.16) | 3.60 (3.00)
Timeline Follow Back [Mean (Standard Deviation); unit: Average days of substance use] — The Timeline Follow Back measures how many days in a specified amount of time, an individual has used an illicit substance. At Baseline, we asked individuals about the past 30 days. The data is noted in average days the substance was consumed.
  Average days of substance use
    Alcohol | 0 (0) | 4.2 (8.84) | 0.2 (0.45) | 1.47 (5.14)
    Cannabis | 6 (12.33) | 0 (0) | 0 (0) | 2 (7.21)
    Crack/Cocaine | 0 (0) | 0.4 (0.89) | 1.4 (1.67) | 0.6 (1.18)
    Amphetamine | 0 (0) | 0 (0) | 0 (0) | 0 (0)
    Opioid Analgesic | 0 (0) | 2.4 (5.37) | 1 (2.24) | 1.13 (3.95)
    Heroin | 0 (0) | 0 (0) | 6.8 (4.1) | 2.27 (3.97)
    Hallucinogen | 0 (0) | 0 (0) | 0 (0) | 0 (0)
    Sedatives | 0 (0) | 0 (0) | 0.2 (0.45) | 0.07 (0.26)
    Benzodiazepines | 0.2 (0.45) | 0 (0) | 0 (0) | 0.07 (0.26)
    Inhalants | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COWS [Mean (Standard Deviation); unit: units on a scale] — The Clinical Opiate Withdrawal Scale (COWS) is an 11-item scale used to help determine the stage or severity of opiate withdrawal and assess the level of physical dependence on opioids. This tool can be used in both inpatient and outpatient settings. This scale has 11 questions with potential scores ranging from 0-48. Lower scores represent less severe opiate withdrawal symptoms and higher scores represent more severe symptoms.
  units on a scale | 0.4 (0.55) | 0.8 (0.84) | 1.6 (1.52) | .93 (1.19)
Positive and Negative Affect Schedule [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Affect Schedule (PANAS) measures positive and negative affect in participants in how they engage with their every day life. This scale consists of 20 questions, 10 measure positive affect and 10 measure negative. Each runs on a scale from 10 to 50. Higher scores indicate higher levels of positive/negative effect and lower scores indicate lower levels.
  units on a scale
    Positive PANAS | 26.2 (9.96) | 31 (3) | 22.2 (2.59) | 26.47 (6.83)
    Negative PANAS | 24.8 (10.64) | 16.6 (2.79) | 21.6 (7.80) | 21.67 (7.98)
Opioid Cravings [Mean (Standard Deviation); unit: units on a scale] — The Opioid Craving scale is based off the validated craving scale by McHugh and colleagues (2021). Answers are on a 10-point scale where 0 represents lower symptoms of opioid cravings and 10 represents high symptoms of opioid cravings.
  units on a scale | 1.2 (1.30) | 2.4 (3.29) | 8.2 (1.48) | 3.31 (3.66)
Timeline Follow Back Alcohol Drinks [Mean (Standard Deviation); unit: numbers of drinks per drinking day] | 0 (0) | 2.05 (0.22) | 2 (0) | 2.05 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cue-reactivity
Description: The primary outcomes is cue-induced cravings (Opioid Craving Scale). This was measured with a single 10-point likert scale asking about cravings, where 0 represented lower levels of craving and 10 indicated higher levels of cravings. This was given at 3 different time points, pre-cue, post-neutral, and post-drug images. Cue-induced craving is the difference between drug cue and pre-cue scores.
Time Frame: Visit 2 and 3 (at least 1 week apart)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cannabidiol 600mg: In this visit, patients received 600mg of Cannabidiol.
  Please note this includes all study visits in which participants received CBD.
- Placebo: In this visit, patients received matching placebo.
  Please note this includes all visits in which participants received placebo.
Arm/Group | Cannabidiol 600mg | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Pre-cue | 0.7 (1.3) | 1.1 (2.0)
  Post-drug cue | 0.9 (1.1) | 2.4 (1.7)
  Post-neutral cue | 0.5 (1.3) | 1.1 (2.0)
  Cue-induced craving | 0.2 (0.79) | 1.3 (1.9)

2. Secondary Outcome: Delayed Discount
Description: Monetary Choice Questionnaire will be used to calculate impulse decision making. This is a 27-item self-administered questionnaire where participants choose between a smaller, immediate monetary reward and a larger, delayed monetary reward. A participants score is between one of the two endpoints (0.25 or 0.00016). If an individual is more likely to prefer the delayed versus immediate reward, their score is more likely to be closer to the 0.00016 endpoint. Please note the rate of delayed discounting is not the same for each question.
Time Frame: Visit 2 and 3 (at least 1 week apart)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cannabidiol 600mg: In this study visit, participants received Cannabidiol 600mg
  This includes all study visits in which participants received CBD.
- Placebo: In this study visit, participants received matched placebo
  Please note this includes all study visits in which participants received placebo.
Arm/Group | Cannabidiol 600mg | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | 0.020 (0.024) | 0.039 (0.075)

3. Secondary Outcome: Decision Making
Description: Iowa Gambling Task will be used to assess impulsive decision-making. The larger the number, the more "safer" options were chosen. This is measured by taking the total number of "risky" choices and subtracting it from the "less risky" choices. The lower the number, the more "high risky" options were chosen. If participants chose the less risky option, they received a positive point, if individuals picked the riskier choice, they received a negative point. Negative values indicate a participant chose more riskier decisions than less-risky, whereas positive values indicate participants chose the less riskier decision more often. The lowest score an individual could receive is -100 (very risk) to 100 (least risky).
Time Frame: Visit 2 and 3 (at least 1 week apart)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cannabidiol 600mg.: In this study visit, all participants received Cannabidiol 600mg.
  Please note this includes all study visits in which participants received CBD.
- Placebo: In this visit, all participants received Placebo.
  Please note this includes all study visits in which participants received placebo.
Arm/Group | Cannabidiol 600mg. | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | 2.2 (9.3) | -6.4 (18.9)

4. Secondary Outcome: Attentional Bias
Description: Visual probe task will be used to assess attentional bias to drug-related cues. Opioid-related and neutral images will be used. Each trial will begin with a fixation point lasting 500ms. A pair of images then will appear on the left and right of the screen for either a short (200ms) or long (500ms) stimulus duration to assess automatic orientating and controlled attention processing, respectively. Image pairs will be replaced by a probe in the location of either the opioid-related or neutral image. The probe will remain until the participant responds to identify the probe orientation by pressing the response keys as quickly as possible. Attentional bias is calculated as the difference in reaction time (RT) between when the probe replaced the neutral compared with the opioid-related images (i.e. RTneutral - RTopioid). Therefore the more positive the number, the less attentional bias toward drug cue, and a negative number represents more attentional bias toward the drug cue.
Time Frame: Visit 2 and 3 (at least 1 week apart)
Measure: Mean (Standard Deviation); unit: miliseconds
Groups:
- Cannabidiol 600mg: In this study visit, all participants received Cannabidiol 600mg.
  Please note this is the combination of all participants' CBD visit.
- Placebo: In this study visit, all participants received placebo.
  Please note this is the combination of all 10 participants' placebo visit.
Arm/Group | Cannabidiol 600mg | Placebo
Number analyzed (Participants) | 10 | 10
miliseconds
  Automatic orienting | -80.4 (298.8) | 100.3 (123.5)
  Controlled attention | 145.2 (392.3) | -93.1 (268.5)

5. Secondary Outcome: Stress-reactivity
Description: Physiologic and subjective stress will be assessed. Stress-reactivity was measured by participants mirror tracing an image on a compute screen where a loud beeping noise would occur if a participant took too long or went outside the lines. It's measured in ms and the longer someone stayed on the task, the better ability they have to react stress.
Time Frame: Visit 2 and 3 (at least 1 week apart)
Measure: Mean (Standard Deviation); unit: miliseconds
Groups:
- Cannabidiol 600mg: Cannabidiol 100 MG/ML [Epidiolex]: 600mg session
- Placebo Session: These results display when all participants received placebo
Arm/Group | Cannabidiol 600mg | Placebo Session
Number analyzed (Participants) | 10 | 10
miliseconds | 59.00 (37.75) | 99.83 (100.78)

6. Secondary Outcome: Stress-Reactivity (Physiological)
Description: For this outcome, participants received a salivary cortisol test prior to, immediately after, and 20 minutes after the cue-reactivity paradigm. Lower levels indicate lower levels of salivary cortisol in the sample.
Time Frame: Visit 2 and 3 (at least 1 week apart)
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Cannabidiol 600mg | Placebo Session
Number analyzed (Participants) | 10 | 10
mcg/dL
  Pre-Paradigm | 0.0855 (0.0579) | 0.1542 (0.179)
  Post-Paradigm | 0.0745 (0.272) | 0.0816 (0.045)
  20 Minutes Post Paradigm | 0.0828 (0.060) | 0.0806 (0.0429)

ADVERSE EVENTS:
Time Frame: 3 weeks - 3 months (participants were enrolled a minimum of 3 weeks and up to 3 months. There was no limit of time between second and third study visit).
Description: Adverse events were monitored and screened for, but no participants reported any adverse events.
Groups:
- Cannabidiol 600mg: All subjects will receive 600mg of oral cannabidiol in a double-blind fashion. Cannabidiol will be provided using Epidiolex™ oral solution 100mg/mL. Following administration, a battery of tests will be conducted to examine reward- and stress-related neurocognitive processes.
  Cannabidiol 100 MG/ML [Epidiolex]: 600mg
  This arm represents the visits all participants received CBD.
- Placebo Arm: Participants will receive a matched placebo the opposite visit they received CBD. Following administration, a battery of tests will be conducted to examine reward- and stress-related neurocognitive processes.
  This arm represents the visits all participants received placebo.
Arm/Group | Cannabidiol 600mg | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT04982029/Prot_SAP_ICF_000.pdf